CLINICAL TRIAL: NCT00238433
Title: A Phase II Study to Evaluate the Safety and Efficacy of IV Busulfan, Melphalan, and Thiotepa (BuMelTT) Followed By Autologous PBSC Infusion for Patients With Hodgkin's Disease and Non-Hodgkin's Lymphoma
Brief Title: Busulfan, Melphalan, and Thiotepa in Treating Patients Who Are Undergoing an Autologous Stem Cell Transplant for Hodgkin's or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard Maziarz, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000248; P30CA069533 (NIH); OHSU-HEM-04083-L; OHSU-IRB-248
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous | interventions — Filgrastim; Busulfan; Melphalan; Thiotepa; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- Filgrastim/Melphalan/Thiotepa (Experimental): Biological/Vaccine: filgrastim
  5mcg/kg intravenous piggyback (IVPB) will be administered beginning on day +5 and continued until absolute neutrophil count (ANC) > 1500 for 2 consecutive days.
  Drug: busulfan
  3.2mg/kg/day for 3 days starting on day -8. Each dose of intravenous busulfan will be mixed in a concentration of 0.54 mg/ml of 0.9% saline and infused over 3 hours.
  Drug: melphalan
  50mg/m2/day/iv, infused over 30 minutes on days -5 and -4. The reconstituted melphalan is diluted in 250cc normal saline to a concentration not greater than 0.4 mg/ml.
  Drug: thiotepa
  250 mg/m2/day/iv on days -3 and -2 Procedure/Surgery: bone marrow ablation with stem cell support
  The transplant therapy should begin within 2 weeks of registration, but no sooner then 30 days after the last dose of chemotherapy.
  Procedure/Surgery: peripheral blood stem cell transplantation
  Performed 36-48 hours following last chemotherapy dose.
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: melphalan; Drug: thiotepa; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — 5mcg/kg IVPB will be administered beginning on day +5 and continued until ANC> 1500 for 2 consecutive days.
Drug: busulfan — 3.2mg/kg/day for 3 days starting on day -8. Each dose of intravenous busulfan will be mixed in a concentration of 0.54 mg/ml of 0.9% saline and infused over 3 hours.
Drug: melphalan — 50mg/m2/day/iv, infused over 30 minutes on days -5 and -4. The reconstituted melphalan is diluted in 250cc normal saline to a concentration not greater than 0.4 mg/ml.
Drug: thiotepa — 250 mg/m2/day/iv on days -3 and -2
Procedure: bone marrow ablation with stem cell support — The transplant therapy should begin within 2 weeks of registration, but no sooner then 30 days after the last dose of chemotherapy.
Procedure: peripheral blood stem cell transplantation — Performed 36-48 hours following last chemotherapy dose.

SUMMARY:
RATIONALE: Chemotherapy, such as busulfan, melphalan, and thiotepa, may destroy cancerous blood-forming cells (stem cells) in the blood and bone marrow. Giving the patient their healthy stem cells will help their bone marrow make new stem cells that become red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well busulfan, melphalan, and thiotepa work in treating patients who are undergoing an autologous stem cell transplant for Hodgkin's or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic efficacy of a myeloablative preparative regimen comprising busulfan, melphalan, and thiotepa followed by autologous peripheral blood stem cell (PBSC) transplantation in patients with Hodgkin's or non-Hodgkin's lymphoma.
* Determine the toxic effects of this preparative regimen in these patients.

OUTLINE:

* Myeloablative preparative regimen: Patients receive busulfan IV over 3 hours on days -8 to -6, melphalan IV over 15-30 minutes on days -5 and -4, and thiotepa IV over 2 hours on days -3 and -2.
* Peripheral blood stem cell (PBSC) transplantation: Patients undergo PBSC transplantation on day 0 followed by filgrastim (G-CSF) IV over 30 minutes beginning on day 5 and continuing until blood counts recover.
* Intrathecal chemotherapy: Patients with a history of treated Central Nervous System (CNS) disease or at high-risk for CNS relapse receive methotrexate and cytarabine intrathecally (IT) for 2 doses each within 10 days prior to transplantation and 4-6 doses each beginning on day 32 post-transplantation.
* Consolidation therapy: Patients with residual bulk disease at 80-100 days post-transplantation that is > 2.5 cm by CT scan may undergo local radiotherapy to residual scar/disease provided it can be encompassed in a single radiation port and the volume of lung to be irradiated is ≤ 20%.

After completion of study treatment, patients are followed weekly for 1 month, monthly for 6 months, every 3 months for 6 months, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Intermediate- or high-grade non-Hodgkin's lymphoma (NHL), meeting 1 of the following criteria:

    * In first complete remission (CR) AND at high-risk for relapse, as defined by all of the following criteria:

      * High age-adjusted International Prognostic Index category AND meets the following criteria at diagnosis:

        * Stage III or IV disease
        * Lactic dehydrogenase abnormal
        * Eastern Cooperative Oncology Group (ECOG) score 0-2
      * Mantle cell histology
    * Primary refractory disease
    * Beyond first CR
  * Low-grade NHL

    * Beyond second relapse
  * Hodgkin's lymphoma

    * Primary refractory disease OR beyond first CR
* Must have an adequate number of stored autologous peripheral blood stem cells (PBSCs) (i.e., 2.0 x 10^6 hematopoietic progenitor cell antigen (CD34)-positive cells/kg)

  * Patients who are not able to mobilize a sufficient number of PBSCs may use bone marrow instead
* No active CNS disease NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 0 to 70

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times ULN

Renal

* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≥ 50 mL/min

Pulmonary

* No significant pulmonary dysfunction, defined as Diffusing Capacity the Lung for Carbon monoxide (DLCO) < 60% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for ≥ 2 months before and during study participation
* HIV negative
* No significant active infection that would preclude PBSC transplantation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior transplantation
* No other concurrent blood products during PBSC transplantation

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* More than 60 days since prior local or regional radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior investigational drugs
* No concurrent amphotericin

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-03; Primary Completion 2015-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Maziarz, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Busulfan/Melphalan/Thiotepa: Treatment:
  Drug: Busulfan 3.2mg/kg/day for 3 days starting on day -8. Each dose of intravenous busulfan will be mixed in a concentration of 0.54 mg/ml of 0.9% saline and infused over 3 hours.
  Drug: Melphalan 50mg/m2/day/iv, infused over 30 minutes on days -5 and -4. The reconstituted melphalan is diluted in 250cc normal saline to a concentration not greater than 0.4 mg/ml.
  Drug: Thiotepa 250 mg/m2/day/iv on days -3 and -2.
  Procedure/Surgery: Peripheral blood stem cell transplantation. Performed 36-48 hours following last chemotherapy dose.
  The transplant therapy should begin within 2 weeks of registration, but no sooner then 30 days after the last dose of chemotherapy.
  Administration Growth Factor: Filgrastim 5mcg/kg intravenous piggyback (IVPB) will be administered beginning on day +5 and continued until absolute neutrophil count (ANC) > 1500 for 2 consecutive days.
Period: Overall Study
Arm/Group | Busulfan/Melphalan/Thiotepa
Started | 37
Completed | 34
Not Completed | 3
Not completed — Screen failure | 1
Not completed — Lost to Follow-up | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Busulfan/Melphalan/Thiotepa: Treatment Plan:
  Drug: Busulfan 3.2mg/kg/day for 3 days starting on day -8. Each dose of intravenous busulfan will be mixed in a concentration of 0.54 mg/ml of 0.9% saline and infused over 3 hours.
  Drug: Melphalan 50mg/m2/day/iv, infused over 30 minutes on days -5 and -4. The reconstituted melphalan is diluted in 250cc normal saline to a concentration not greater than 0.4 mg/ml.
  Drug: Thiotepa 250 mg/m2/day/iv on days -3 and -2.
  Procedure/Surgery: Peripheral blood stem cell transplantation. Performed 36-48 hours following last chemotherapy dose.
  The transplant therapy should begin within 2 weeks of registration, but no sooner then 30 days after the last dose of chemotherapy.
  Administration Growth Factor: Filgrastim 5mcg/kg IVPB will be administered beginning on day +5 and continued until ANC> 1500 for 2 consecutive days.
Arm/Group | Busulfan/Melphalan/Thiotepa
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival
Description: The data presented below represents the total number of subjects (out of 36) that reached disease-free survival status during Months 3, 6, 9, 12, 18, and 24 time points.
Time Frame: 3, 6, 9, 12, 18, and 24 months post transplantation
Measure: Count of Participants; unit: Participants
Groups:
- Busulfan/Melphalan/Thiotepa: Busulfan: 3.2mg/kg/day for 3 days starting on day -8. Each dose of intravenous busulfan will be mixed in a concentration of 0.54 mg/ml of 0.9% saline and infused over 3 hours.
  Melphalan: 50mg/m2/day/iv, infused over 30 minutes on days -5 and -4. The reconstituted melphalan is diluted in 250cc normal saline to a concentration not greater than 0.4 mg/ml.
  Thiotepa: 250 mg/m2/day/iv on days -3 and -2
  Procedure/Surgery: bone marrow ablation with stem cell support
  The transplant therapy should begin within 2 weeks of registration, but no sooner then 30 days after the last dose of chemotherapy.
  Procedure/Surgery: Peripheral blood stem cell transplantation. Performed 36-48 hours following last chemotherapy dose.
  Growth factor administration: Filgrastim 5mcg/kg IVPB will be administered beginning on day +5 and continued until ANC> 1500 for 2 consecutive days.
Arm/Group | Busulfan/Melphalan/Thiotepa
Number analyzed (Participants) | 36
Participants
  3 months | 34
  6 months | 30
  9 months | 28
  12 months | 25
  18 months | 24
  24 months | 22

2. Primary Outcome: Therapy-Related Toxicities
Description: The table presented below reflects how many participants (out of 36 total) presented an adverse event related to the treatment regimen within each toxicity category. To review specific adverse events, both related and unrelated to study treatment, please refer to Adverse Events Section.
Time Frame: Through 24 months post transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Busulfan/Melphalan/Thiotepa
Number analyzed (Participants) | 36
Participants
  Dermatological Toxicities | 3
  Gastrointestinal Toxicities | 26
  Immune System Toxicites | 1
  Infections | 33
  Metabolic Toxicities | 3
  Respiratory Toxicities | 2
  Vascular Toxicities | 1

ADVERSE EVENTS:
Time Frame: For all adverse events grade 3 or higher is recorded for the first 100 days post transplant. After 100 days post transplant, all unexpected grade 3 and 4 adverse events will be recorded and reported.
Groups:
- BuMelTT: *For all adverse events grade 3 or higher is recorded for the first 100 days post transplant. After 100 days post transplant, all unexpected grade 3 and 4 adverse events will be recorded and reported.
  TREATMENT PLAN:
  Busulfan: 3.2mg/kg/day for 3 days starting on day -8. Each dose of intravenous busulfan will be mixed in a concentration of 0.54 mg/ml of 0.9% saline and infused over 3 hours.
  Melphalan: 50mg/m2/day/iv, infused over 30 minutes on days -5 and -4. The reconstituted melphalan is diluted in 250cc normal saline to a concentration not greater than 0.4 mg/ml.
  Thiotepa: 250 mg/m2/day/iv on days -3 and -2
  Procedure/Surgery: bone marrow ablation with stem cell support
  The transplant therapy should begin within 2 weeks of registration, but no sooner then 30 days after the last dose of chemotherapy.
  Procedure/Surgery: Peripheral blood stem cell transplantation. Performed 36-48 hours following last chemotherapy dose.
  Growth factor administration: Filgrastim
Arm/Group | BuMelTT
Serious Adverse Events (participants affected / at risk) | 36/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BuMelTT (N=36)
Cardiac arrest (Cardiac disorders) | 1 — Unrelated to treatment regimen.
Abdominal pain (Gastrointestinal disorders) | 1 — Related to treatment regimen.
Anorexia (Gastrointestinal disorders) | 5 — Related to treatment regimen.
Colonic obstruction (Gastrointestinal disorders) | 1 — Unrelated to treatment regimen.
Dehydration (Gastrointestinal disorders) | 1 — Related to treatment regimen.
Ileum obstruction (Gastrointestinal disorders) | 1 — Related to treatment regimen.
Mucositis (Gastrointestinal disorders) | 20 — Related to treatment regimen.
Nausea (Gastrointestinal disorders) | 8 — Related to treatment regimen.
Vomiting (Gastrointestinal disorders) | 2 — Related to treatment regimen.
Febrile neutropenia (Infections and infestations) | 33 — Related to treatment regimen.
Influenza A (Infections and infestations) | 1 — Unrelated to treatment regimen.
Sepsis (Infections and infestations) | 2 — Related to treatment regimen.
Vasovagal reaction (Nervous system disorders) | 1 — Unrelated to treatment regimen.
Opioid overdose (Psychiatric disorders) | 1 — Unrelated to treatment regimen.
Suicide attempt (Psychiatric disorders) | 1 — Unrelated to treatment regimen.
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 — Unrelated to treatment regimen.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 — Unrelated to treatment regimen.
Hypotension (Vascular disorders) | 1 — Related to treatment regimen.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BuMelTT (N=36)
Constipation (Gastrointestinal disorders) | 1 — Unrelated to treatment regimen.
Diarrhea (Gastrointestinal disorders) | 5 — Related to treatment regimen.
Distended abdomen (Gastrointestinal disorders) | 1 — Unrelated to treatment regimen.
Esophagitis (Gastrointestinal disorders) | 1 — Related to treatment regimen.
Fatigue (General disorders) | 2 — Unrelated to treatment regimen.
Auto GVHD (Immune system disorders) | 1 — Related to treatment regimen.
Clostridium difficile colitis (C. diff) (Infections and infestations) | 1 — Unrelated to treatment regimen.
Entercolitis (Infections and infestations) | 1 — Related to treatment regimen.
Pancolitis (Infections and infestations) | 1 — Related to treatment regimen.
Abnormal ALT (alanine aminotransferase ) lab result (Metabolism and nutrition disorders) | 1 — Unrelated to treatment regimen.
Abnormal amylase lab result (Metabolism and nutrition disorders) | 1 — Unrelated to treatment regimen.
Hyperglycemia (Metabolism and nutrition disorders) | 1 — Unrelated to treatment regimen.
Hyperkalemia (Metabolism and nutrition disorders) | 1 — Unrelated to treatment regimen.
Hypermagnesemia (Metabolism and nutrition disorders) | 1 — Unrelated to treatment regimen.
Hyperuricemia (Metabolism and nutrition disorders) | 1 — Unrelated to treatment regimen.
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 — Related to treatment regimen.
Hypocalcemia (Metabolism and nutrition disorders) | 1 — Unrelated to treatment regimen.
Hypokalemia (Metabolism and nutrition disorders) | 9 — Unrelated to treatment regimen.
Hyponatremia (Metabolism and nutrition disorders) | 5 — Unrelated to treatment regimen.
Hypophosphatemia (Metabolism and nutrition disorders) | 14 — Unrelated to treatment regimen.
Muscle weakness (lower limb) (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to treatment regimen.
Eating disorder (Psychiatric disorders) | 1 — Unrelated to treatment regimen.
Urinary frequency/urgency (Renal and urinary disorders) | 1 — Unrelated to treatment regimen.
Urinary retention (Renal and urinary disorders) | 1 — Unrelated to treatment regimen.
Bronchitis/early bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 — Related to treatment regimen.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 — Unrelated to treatment regimen.
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 — Related to treatment regimen.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 — Unrelated to treatment regimen.
General skin rash (Skin and subcutaneous tissue disorders) | 1 — Unrelated to treatment regimen.
Thiotepa-induced skin rash (Skin and subcutaneous tissue disorders) | 3 — Related to treatment regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes